CLINICAL TRIAL: NCT03046238
Title: Efficacy and Safety of Dexmedetomidine Added to Modified Pectoral's Block in Patient Undergoing Breast Cancer Surgery :A Comparative Study
Brief Title: Efficacy and Safety of Dexmedetomidine Added to Modified Pectoral's Block in Breast Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Dr.mohamad farouk mohamad, lecturer of anesthesia,ICU and pain relief, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 222
Record Dates: First submitted 2017-02-02; First posted 2017-02-08 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer Patients
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dexmetedomedine (Active Comparator): preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine plus Dexmedetomidine (1 µg/kg)
  Interventions: Drug: Dexmedetomidine
- control (Placebo Comparator): preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexmedetomidine — preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine plus Dexmedetomidine (1 µg/kg)
  Arms: dexmetedomedine
Drug: placebo — preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine
  Other Names: control
  Arms: control

SUMMARY:
To Evaluate the effect of addition of Dexmedetomedine to ultrasound guided modified Pecs block on post operative analgesia & stress response in patient undergoing modified radical mastectomy.

DETAILED DESCRIPTION:
60 patients (age ≥29 years) who scheduled for modified radical mastectomy surgery under general anesthesia. Group I (Bupivacaine group): patients underwent modified radical mastectomy were given preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine divided into 10 ml injected between the pectoralis muscles on the interfasial plane, and 20 ml injected between the Pectoralis minor muscle and the serratus muscle.Group II (Bupivacaine + Dexmedetomidine group) : preoperative ultrasound guided modified Pecs block with 30 mL of 0.25% bupivacaine plus Dexmedetomidine (1 µg/kg) divided into 20 ml injected between the pectoralis muscles on the interfasial plane , and 10 ml injected between the Pectoralis minor muscle and the serratus muscle.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II patients
* weight 50- 100 kg)

Exclusion Criteria:

* a history of bleeding diathesis,
* relevant drug allergy
* opioid dependence,
* sepsis,
* those with psychiatric illnesses

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-04-02 (Estimated); Study Completion 2017-04-02 (Estimated)

PRIMARY OUTCOMES:
morphine consumption mg/day | 48 HOURS
  by Patient-controlled analgesia (PCA) device
Visual Analog Scale (VAS), scored from 0-10 | 48 hours
  pain measurement

SECONDARY OUTCOMES:
first request of analgesia | 48 hours
  time of the first request of analgesia postoperative if the VAS ≥ 3
level of stress hormones | 48 hours
  cortisol level
Adverse Events | 48 hours
  Nausea Vomiting Bradycardia Hypotension Arrhythmia Pneumothorax Vascular injury Nausea Vomiting Bradycardia Hypotension Arrhythmia Pneumothorax Vascular injury Nausea,Vomiting,Arrhythmia.Hypotension,Pneumothorax,Vascular injury andItching

CONTACTS AND LOCATIONS:
Overall Officials: mohamad F mohamad, MD, Principal Investigator — Assiut University; Saher mohamad, MD, Study Director — Cancer Institute, Anesthesia, Intensive Care, and Pain Management, South Egypt Cancer Institute, Assiut University, Assiut, Egypt.
Locations (1):
- South Egypt Cancer Institute, Assiut University, Assiut, Egypt., Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes